CLINICAL TRIAL: NCT07407725
Title: Development of a Clinical Outcome Assessment for Assistive Technologies and Brain-Computer-Interfaces
Brief Title: Clinical Outcome Assessment for AT & BCI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shirley Ryan AbilityLab (Other)
Collaborators: Neuralink Corp (Industry)
Responsible Party: Principal Investigator, Arun Jayaraman, PT, PhD, Director, Max Nader Center for Rehabilitation Technologies & Outcomes Research, Shirley Ryan AbilityLab
Allocation: Not Applicable | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: STU00224714
Record Dates: First submitted 2026-01-22; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Spinal Cord Injury; ALS (Amyotrophic Lateral Sclerosis)
Keywords: iBCI; Brain Computer Interface; Assistive Technology; Clinical Outcome Assessment; dADL; digital activities of daily living
MeSH Terms: conditions — Spinal Cord Injuries; Amyotrophic Lateral Sclerosis | interventions — Electroencephalography

STUDY DESIGN:
Intervention Model Description: Participants will complete the assessment with up to four different devices, and any existing device or iBCI they use in their daily life. It is a randomized, within-subject crossover interventional study in which participants complete standardized digital tasks using multiple assistive technologies in randomized order. There is one arm per technology within each participant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AT/BCI User (Experimental): Participants in this arm will undergo training and a digital assessment using 3 assistive technologies (eye tracker, mouth-operated joystick, non-invasive electroencephalogram (EEG) headset), brain-computer-interfaces, and applicable personal ATs. Participants will experience each of these devices in a randomized order. Participants in this arm will include individuals with a diagnosis of amyotrophic lateral sclerosis (ALS), spinal cord injury (SCI), or healthy individuals.
  Interventions: Device: Eye Tracker; Device: Mouth Operated Joystick; Device: Non-invasive electroencephalogram (EEG) Headset; Device: Implantable Brain-Computer-Interface; Device: Personal Assistive Technology

INTERVENTIONS:
Device: Eye Tracker — The intervention consists of two 40-minute training sessions using a customized Digital Training Interface to practice motor primitives for digital activities (clicking, typing, scrolling, drawing). The first session includes an orientation to the eye-tracking device, calibration, and setup adjustments, after which the clinician will confirm feasibility. Training begins with a guided tutorial followed by eight practice levels, each lasting 3 minutes or until 20 correct targets are achieved. Participants are encouraged to complete all levels and focus on challenging primitives. In-clinic and at-home sessions are scheduled on separate days, with a rest period for in-clinic visits, ensuring adequate rest and retention of learned skills.
  Other Names: Tobii Dynavox PCEye 5
Device: Mouth Operated Joystick — The intervention consists of two 40-minute training sessions using a customized Digital Training Interface to practice motor primitives for digital activities (clicking, typing, scrolling, drawing). The first session includes an orientation to the mouth-operated joystick device, calibration, and setup adjustments, after which the clinician will confirm feasibility. Training begins with a guided tutorial followed by eight practice levels, each lasting 3 minutes or until 20 correct targets are achieved. Participants are encouraged to complete all levels and focus on challenging primitives. In-clinic and at-home sessions are scheduled on separate days, with a rest period for in-clinic visits, ensuring adequate rest and retention of learned skills.
  Other Names: Jouse+
Device: Non-invasive electroencephalogram (EEG) Headset — The intervention consists of two 40-minute training sessions using a customized Digital Training Interface to practice motor primitives for digital activities (clicking, typing, scrolling, drawing). The first session includes an orientation to the non-invasive EEG headset device, calibration, and setup adjustments, after which the clinician will confirm feasibility. Training begins with a guided tutorial followed by eight practice levels, each lasting 3 minutes or until 20 correct targets are achieved. Participants are encouraged to complete all levels and focus on challenging primitives. In-clinic and at-home sessions are scheduled on separate days, with a rest period for in-clinic visits, ensuring adequate rest and retention of learned skills.
  Other Names: EMOTIVE EPOC X
Device: Implantable Brain-Computer-Interface — Participants with an invasive Brain Computer Interface (BCI) implant, primarily recruited via Neuralink, will use the Neuralink N1 or any other implanted BCI. The intervention consists of one 40-minute training session using a customized Digital Training Interface to practice motor primitives for digital activities (clicking, typing, scrolling, drawing). The session begins with setup assistance and calibration to ensure proper positioning. Training includes a guided tutorial followed by eight practice levels, each lasting 3 minutes or until 20 correct targets are achieved. Participants are encouraged to complete all levels and focus on the most challenging primitives. Prior experience with the device justifies the single-session design.
  Other Names: Neuralink N1 Implant
Device: Personal Assistive Technology — Participants already using a personal assistive technology device will complete one 40-minute training session with a customized Digital Training Interface to practice motor primitives for digital activities (clicking, typing, scrolling, drawing). The session begins with setup assistance and positioning. Training includes a guided tutorial followed by eight practice levels, each lasting 3 minutes or until 20 correct targets are achieved. Participants are encouraged to complete all levels and focus on the most challenging primitives. Since the device is already familiar, only a single session is required.

SUMMARY:
Many individuals with severe motor impairments rely on Assistive Technologies (ATs) or Brain-Computer Interfaces (BCIs) to interact with digital devices such as their computers. Clinicians and researchers currently lack a common framework to objectively quantify how much a given AT or BCI improves real-world function or to compare across tools. This project seeks to address this gap by developing a standardized method to objectively assess or compare the functional benefit of these tools on digital independence, i.e., the ability to independently operate computers, phones, and other digital systems, by creating a unique Digital Assessment Interface (DAI).

This assessment will be a simulation of online and digital activities that prior work has determined is important to functional daily living in the digital domain. Participants will complete this assessment with various ATs and BCIs, and these scores will be used to create an index, which will be comprised of performance outcomes, clinician-reported outcomes, and patient-reported outcomes.

The tool aims to quantify and compare digital task performance across devices and user populations. The primary objective of this study is to develop an index. The index will quantify functional performance of individuals using various ATs and BCIs. The secondary objectives are to extensively evaluate the psychometric properties of the index, such as the validity, responsiveness, reliability, and floor/ceiling effects both globally and across different devices and impairment levels, ensuring that it can reliably measure the impact of an AT or BCI on a user's ability to independently operate digital systems; and to characterize the familiarization and use of specific BCI and AT systems with reference to a normative healthy control population.

ELIGIBILITY:
Enrollment will involve three different cohorts, namely a cohort of healthy participant, a cohort of ALS/SCI participant who underwent the implant of an invasive BCI device, and a cohort of ALS/SCI participants without any implanted BCI device.

Below are listed the inclusion and exclusion criteria for each diagnostic group.

Spinal Cord Injury (SCI):

Inclusion Criteria:

* Age at or above 18 years old;
* Diagnosis of spinal cord injury, at the level of T1 or above levels (between C1 and T1);
* Ability to communicate independently or with a support device, or with a legal representative;
* Ability to participate in a study session for about 3 hours (e.g., endurance, fatigue), which may include breaks as needed.

Exclusion Criteria:

* Participation in another trial that would conflict with the current study or clinical endpoint interference may occur.

Amyotrophic Lateral Sclerosis (ALS):

Inclusion criteria:

* Age at or above 18 years old;
* Diagnosis of amyotrophic lateral sclerosis;
* Ability to communicate independently, with a support device, or with a legal representative;
* Ability to participate in a study session for about 3 hours (e.g., endurance, fatigue), which may include breaks as needed.

Exclusion criteria:

● Participation in another trial that would conflict with the current study or clinical endpoint interference may occur.

Healthy Controls:

Inclusion criteria:

* Age at or above 18 years old;
* No history of neurological or psychiatric disorders;
* Ability to provide written informed consent;
* Ability to participate in a study session for about 3 hours (e.g., endurance, fatigue), which may include breaks as needed.

Exclusion criteria:

* Participation in another trial that would conflict with the current study or clinical endpoint interference may occur;
* Cognitive, visual, or auditory deficits that would interfere with study participation;
* Current or prior diagnosis or condition that could confound study assessments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01-08 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Performance Outcomes (PerfOs) | Through study completion, every visit during the Digital Assessment Interface.
  Quantitative metrics will be extracted from a customized Digital Assessment Interface simulating digital activities of daily living (dADLs, e.g., online shopping, texting, gaming, booking appointments). Metrics will be collected for each motor primitive (clicking, scrolling, typing, click-and-drag) to evaluate performance, including click accuracy, time to target, number of errors, cursor trajectory, words per minute, and percentage of correct letters/characters.
Demographics and Medical Intake Questionnaire | Day 1
  Demographic characteristics such as age and sex will be considered for index development (primary objective), along with level of education and race/ethnicity for index validation and characterization of Assistive Technology/Brain Computer Interface systems (secondary objective). Medical intake information, including diagnosis, will be considered for index development (primary), validation (secondary), and device characterization (secondary).
NASA Task Load Index | Through study completion, every visit after an attempt or completion of the Digital Assessment Interface.
  A self-report questionnaire for measuring the perceived workload of the use of each assistive technology across 6 domains: mental demand, physical demand, temporal demand, performance, effort, and frustration. This will be conducted to inform index development (primary objective) as well as validation and device characterization (secondary objectives).
NASA Task Load Index - Clinician's perspective | Through study completion, every visit after an attempt or completion of the Digital Assessment Interface.
  A self-report questionnaire for measuring the perceived workload of the use of each assistive technology across 6 domains: mental demand, physical demand, temporal demand, performance, effort, and frustration. This will be conducted as a clinician-reported outcome, where the clinician will evaluate the participant's level of fatigue in performing digital activities of daily living. This measure will be used to inform index development (primary objective) as well as validation and device characterization (secondary objectives).
System Usability Scale (SUS) | Through study completion, every visit after an attempt or completion of the Digital Assessment Interface.
  A brief 10-item questionnaire that measures a system's overall perceived usability. Items are rated on a 5-point Likert scale to measure ease of use, complexity, and user experience. This will be conducted as an outcome measure for index development (primary objective) as well as validation and device characterization (secondary objectives).
System Usability Scale (SUS) - Clinician's perspective | Through study completion, every visit after an attempt or completion of the Digital Assessment Interface.
  A brief 10-item questionnaire that measures a system's overall perceived usability. Items are rated on a 5-point Likert scale to measure ease of use, complexity, and user experience. This will be conducted as a clinician-reported outcome, where the clinician will evaluate the participant's usability of the experimental device in performing digital activities of daily living. This measure will be used to inform index development (primary objective) as well as validation and device characterization (secondary objectives).
Qualitative Questionnaire | Through study completion, every visit after an attempt or completion of the Digital Assessment Interface.
  Modified version of the Canadian Occupational Performance Measure (COPM) to better capture functional digital independence. The qualitative questionnaire is conducted via a semi-structured interview to help participants identify goals in the area of digital independence and rate their performance and satisfaction on a scale. This measure will be used to inform index development (primary objective) as well as validation and device characterization (secondary objectives).
Psychosocial Impact of Assistive Devices (PIAD) | Through study completion, every visit after an attempt or completion of the Digital Assessment Interface
  Self-report questionnaire designed to measure the effects of an assistive device on functional independence, well-being, and quality of life. It is a patient-reported outcome measure that assesses perceptions of competence, adaptability, and self-esteem, helping to understand the user's experience and predict device adoption/abandonment. This measure will be used to inform index development (primary objective) as well as validation and device characterization (secondary objectives).

SECONDARY OUTCOMES:
International Standards for Neurological Classification of Spinal Cord Injury (ISNCSCI) | Day 1
  Classification of motor and sensory impairments that result from a spinal cord injury. This study involves an abbreviated version of the ISNCSCI in the medical intake questionnaire to include C1-T1 sensation, upper extremity and lower extremity motor scores, and a sacral sparing gathered through a short questionnaire. These scores will be translated into a modified ASIA (American Spinal Injury Association Impairment Scale) score for use in the characterization of AT/BCI systems (secondary objective).
Amyotrophic Lateral Sclerosis Functional Rating Scale-Revised (ALSFRS-R) | Day 1
  This scale, as part of the medical intake questionnaire, measures activities of daily living and global function for patients with ALS. The ALSFRS-R provides an estimate of a patient's degree of functional impairment, which can be evaluated serially to objectively assess any response to treatment or progression of disease. This will be utilized in the characterization of the Assistive Technology/Brain Computer Interface systems (secondary objective).
Clinical Evaluation | Day 1
  Components of the clinical evaluation, such as comfort level with an Assistive Technology device and the use and experience with other Assistive Technology devices will be factored into the characterization of the Assistive Technology/Brain Computer Interface systems (secondary objective).
Inpatient Rehabilitation Facility Patient Assessment Instrument (IRF-PAI) Section GG | Day 1
  Standardized evaluation of functional abilities and goals related to self-care and mobility. This assessment provides detailed item-level information on patient function, using a 6-point scale to rate the level of assistance required for various activities, and will be used in the validation of the index and in the characterization of the Assistive Technology/Brain Computer Interface systems (secondary objectives).
Edinburgh Cognitive and Behavioral ALS Screen (ECAS) | Day 1
  Comprehensive screening tool for cognitive and behavioral changes in individuals with amyotrophic lateral sclerosis, which will enable the study team to screen for cognitive changes that may impact study participation and inform Assistive Technology/Brain Computer Interface characterization (secondary objective).
World Health Organization Quality of Life-BREF (WHOQOL-BREF) | Day 1
  Self-report questionnaire that addresses 4 quality of life domains: physical health, psychological health, social relationships, and environment. 2 other items measure overall quality of life and general health. This patient-reported outcome will be used in the validation of the index and in the characterization of the Assistive Technology/Brain Computer Interface systems (secondary objectives).

CONTACTS AND LOCATIONS:
Locations (1):
- Shirley Ryan AbilityLab, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sawyer A, Brannigan J, Spielman L; BCI Functional Outcome Measures Group; Putrino D, Fry A. Development of a novel clinical outcome assessment: digital instrumental activities of daily living. EBioMedicine. 2025 Jun;116:105732. doi: 10.1016/j.ebiom.2025.105732. Epub 2025 May 26. PMID 40424668
- [Background] Consortium for Spinal Cord Medicine. Outcomes following traumatic spinal cord injury: clinical practice guidelines for health-care professionals. J Spinal Cord Med. 2000 Winter;23(4):289-316. doi: 10.1080/10790268.2000.11753539. No abstract available. PMID 17536300
- [Background] Anderson K, Aito S, Atkins M, Biering-Sorensen F, Charlifue S, Curt A, Ditunno J, Glass C, Marino R, Marshall R, Mulcahey MJ, Post M, Savic G, Scivoletto G, Catz A; Functional Recovery Outcome Measures Work Group. Functional recovery measures for spinal cord injury: an evidence-based review for clinical practice and research. J Spinal Cord Med. 2008;31(2):133-44. doi: 10.1080/10790268.2008.11760704. PMID 18581660
- [Background] Pupillo E, Messina P, Giussani G, Logroscino G, Zoccolella S, Chio A, Calvo A, Corbo M, Lunetta C, Marin B, Mitchell D, Hardiman O, Rooney J, Stevic Z, Bandettini di Poggio M, Filosto M, Cotelli MS, Perini M, Riva N, Tremolizzo L, Vitelli E, Damiani D, Beghi E; EURALS Consortium. Physical activity and amyotrophic lateral sclerosis: a European population-based case-control study. Ann Neurol. 2014 May;75(5):708-16. doi: 10.1002/ana.24150. Epub 2014 May 21. PMID 24706338
- [Background] Turner MR, Hardiman O, Benatar M, Brooks BR, Chio A, de Carvalho M, Ince PG, Lin C, Miller RG, Mitsumoto H, Nicholson G, Ravits J, Shaw PJ, Swash M, Talbot K, Traynor BJ, Van den Berg LH, Veldink JH, Vucic S, Kiernan MC. Controversies and priorities in amyotrophic lateral sclerosis. Lancet Neurol. 2013 Mar;12(3):310-22. doi: 10.1016/S1474-4422(13)70036-X. PMID 23415570
- [Background] Anderson KD. Targeting recovery: priorities of the spinal cord-injured population. J Neurotrauma. 2004 Oct;21(10):1371-83. doi: 10.1089/neu.2004.21.1371. PMID 15672628
- [Background] van Middendorp JJ, Hosman AJ, Donders AR, Pouw MH, Ditunno JF Jr, Curt A, Geurts AC, Van de Meent H; EM-SCI Study Group. A clinical prediction rule for ambulation outcomes after traumatic spinal cord injury: a longitudinal cohort study. Lancet. 2011 Mar 19;377(9770):1004-10. doi: 10.1016/S0140-6736(10)62276-3. Epub 2011 Mar 4. PMID 21377202
- [Background] Fessler EB, Brown RT, Miller RK. Rebooting Instrumental Activities of Daily Living for the 21st Century. Ann Intern Med. 2022 Feb;175(2):278-279. doi: 10.7326/M21-3065. Epub 2021 Dec 21. No abstract available. PMID 34928697
- [Background] Lu X, Yao Y, Jin Y. Digital exclusion and functional dependence in older people: Findings from five longitudinal cohort studies. EClinicalMedicine. 2022 Oct 31;54:101708. doi: 10.1016/j.eclinm.2022.101708. eCollection 2022 Dec. PMID 36353265
- [Background] Mois G, Rogers WA. Developing a Framework for Digital Activities of Daily Living. Gerontologist. 2024 Oct 1;64(10):gnae110. doi: 10.1093/geront/gnae110. PMID 39163564
- [Background] Rigby P, Ryan SE, Campbell KA. Electronic aids to daily living and quality of life for persons with tetraplegia. Disabil Rehabil Assist Technol. 2011;6(3):260-7. doi: 10.3109/17483107.2010.522678. Epub 2010 Oct 1. PMID 20883120
- [Background] Fairman, A. D., Indradhirmaya, F. A., Osal, R. B. & Saptono, A. Iterative User-Centered Design of the Mobile Device Assessment Tool (MoDAT). Technologies 13, 358 (2025).
- [Background] Dohle, E. et al. Outcome measures in implantable brain-computer interface research: a systematic review. 2024.10.15.24315534 Preprint at https://doi.org/10.1101/2024.10.15.24315534 (2024).
- [Background] Roberts TT, Leonard GR, Cepela DJ. Classifications In Brief: American Spinal Injury Association (ASIA) Impairment Scale. Clin Orthop Relat Res. 2017 May;475(5):1499-1504. doi: 10.1007/s11999-016-5133-4. Epub 2016 Nov 4. No abstract available. PMID 27815685
- [Background] Cedarbaum JM, Stambler N, Malta E, Fuller C, Hilt D, Thurmond B, Nakanishi A. The ALSFRS-R: a revised ALS functional rating scale that incorporates assessments of respiratory function. BDNF ALS Study Group (Phase III). J Neurol Sci. 1999 Oct 31;169(1-2):13-21. doi: 10.1016/s0022-510x(99)00210-5. PMID 10540002
- [Background] Huang TT, Wang WS. Comparison of three established measures of fear of falling in community-dwelling older adults: psychometric testing. Int J Nurs Stud. 2009 Oct;46(10):1313-9. doi: 10.1016/j.ijnurstu.2009.03.010. Epub 2009 Apr 24. PMID 19394017
- [Background] Kalsi-Ryan S, Chan C, Verrier M, Curt A, Fehlings M, Bolliger M, Velstra IM; GRASSP Cross Sectional Study Team; GRASSP Longitudinal Study Team. The graded redefined assessment of strength sensibility and prehension version 2 (GV2): Psychometric properties. J Spinal Cord Med. 2019 Oct;42(sup1):149-157. doi: 10.1080/10790268.2019.1616950. PMID 31573454
- [Background] Crockford CJ, Kleynhans M, Wilton E, Radakovic R, Newton J, Niven EH, Al-Chalabi A, Hardiman O, Bak TH, Abrahams S. ECAS A-B-C: alternate forms of the Edinburgh Cognitive and Behavioural ALS Screen. Amyotroph Lateral Scler Frontotemporal Degener. 2018 Feb;19(1-2):57-64. doi: 10.1080/21678421.2017.1407793. Epub 2017 Dec 5. PMID 29205065
- [Background] Jordan, P.W., Thomas, B., McClelland, I.L., & Weerdmeester, B. (Eds.). (1996). Usability Evaluation In Industry (1st ed.). CRC Press. https://doi.org/10.1201/9781498710411
- [Background] Hart, S. G. & Staveland, L. E. Development of NASA-TLX (Task Load Index): Results of Empirical and Theoretical Research. in Advances in Psychology (eds Hancock, P. A. & Meshkati, N.) vol. 52 139-183 (North-Holland, 1988).
- [Background] Eyssen IC, Beelen A, Dedding C, Cardol M, Dekker J. The reproducibility of the Canadian Occupational Performance Measure. Clin Rehabil. 2005 Dec;19(8):888-94. doi: 10.1191/0269215505cr883oa. PMID 16323388
- [Background] Saeed SS, Hejazi-Shirmard M, Akbarzadeh Baghban A, Jutai J, Rezaee M. Translation and validation of the Persian version of "The Psychosocial Impact of Assistive Devices Scale" in patients with neurological disorders. Assist Technol. 2025 Feb 14;37(sup1):S125-S130. doi: 10.1080/10400435.2024.2363383. Epub 2024 Jun 25. PMID 38916516
- [Background] Deutsch A, Palmer L, Vaughan M, McMullen T, Kwon S, Karmarkar A, Ingber MJ. Reliability and Validity of the Inpatient Rehabilitation Facility Discharge Mobility and Self-Care Quality Measures. J Am Med Dir Assoc. 2023 May;24(5):723-728.e4. doi: 10.1016/j.jamda.2023.03.015. Epub 2023 Apr 5. PMID 37030324
- See also: WHO- Global report on assistive technology — http://www.who.int/publications/i/item/9789240049451
- See also: CMS- IRF-PAI Section GG — http://www.cms.gov/medicare/quality/inpatient-rehabilitation-facility/irf-pai-and-irf-qrp-manual